CLINICAL TRIAL: NCT04775056
Title: A Study to Describe the Safety, Tolerability, Immunogenicity, and Efficacy of Vaccines Against COVID-19 in the Real World
Brief Title: A Study to Evaluate Vaccines Against COVID-19 in the Real World
Status: Withdrawn | Type: Observational
Why Stopped: No sponsor
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Other Study IDs: APASL_COVID-19 Vaccine_Ab
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Liver Disease; Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection and the resulting coronavirus disease 2019 (COVID-19) have afflicted tens of millions of people in a worldwide pandemic. Considering its high mortality and rapid spread, an effective vaccine is urgently needed to control this pandemic. Recently, mass vaccination campaigns using newly approved vaccines, ranging from conventional viral and protein-based vaccines to those that are more cutting edge, including DNA- and mRNA-based vaccines are beginning in many parts of the world. Randomized clinical trials of different vaccines reported efficacies for preventing COVID-19 in the range of 50% to 95%.

Although these randomized clinical trials are considered the "gold standard" for evaluating intervention effects, they have notable limitations of sample size and subgroup analysis, restrictive inclusion criteria, and a highly controlled setting that may not be replicated in a mass vaccine rollout.

The aim of this study is to evaluate the safety, tolerability, immunogenicity, and efficacy of different vaccines against COVID-19 under real-world practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects received COVID-19 vaccines;
* Able to comprehend and provide written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* Not received any COVID-19 vaccines;
* Not willing to participate and/or give their written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who received COVID-19 vaccines under real-life practice conditions in the World
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-seroconversion rates of neutralizing antibody | The 4 weeks after the second dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4 fold increase from baseline.

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-28 after each dose vaccination
  Incidence of adverse reactions after each dose vaccination
Immunogenicity index-seropositive rates of neutralizing antibody | The 4, 12, 24, and 48 weeks after the second dose vaccination
  neutralizing antibody assay will be performed using the micro-neutralization method, and subjects with a antibody titer ≥1:8 will defined as seropositive.

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity & Health Medical Group
Locations (1):
- Humanity & Health Medical Group, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No